CLINICAL TRIAL: NCT00065104
Title: Dehydroepiandrosterone Effects on HIV-1 Replication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000512-01 (NIH); AbramsD
Record Dates: First submitted 2003-07-17; First posted 2003-07-18 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections
Keywords: HIV; DHEA; immune system; hormones; body composition; quality of life
MeSH Terms: conditions — HIV Infections | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: DHEA

SUMMARY:
This study's purpose is to learn how dehydroepiandrosterone (DHEA) affects the HIV virus, the immune system, hormone levels, body composition and quality of life.

ELIGIBILITY:
Inclusion criteria:

* Evidence of HIV-1 infection
* HIV RNA <50 copies/mL
* Stable antiretroviral treatment regimen for at least 8 weeks
* Age 18 years or older
* Normal pap smear and mammograph within 1 year (females)
* Normal prostate-specific antigen level with in one year, age adjusted (males)

Exclusion criteria:

* Active opportunistic infections or malignancy other than localized cutaneous KS lesions
* Concurrent or prior use within the past 8 weeks of DHA, testosterone, other anabolic steroids, corticosteroids, megestrol acetate, growth hormone, IL-2, or thalidomide
* Diagnosis of AIDS Dementia Complex (stage II or higher)
* Active substance abuse (e.g., alcohol or injection drugs)
* Evidence of severe liver dysfunction or hepatic transaminases greater than 3x the upper normal limit
* Pregnant or breast-feeding
* History of endocrinologically-responsive tumors (e.g., breast, ovarian, uterine, or prostatic cancer, or malignant melanoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2000-10; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- Community Consortium, San Francisco, California, United States